CLINICAL TRIAL: NCT03181919
Title: Letrozole Step-up Protocol for Ovulation Induction in Infertile Women With PCOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Dr. Abou Bakr Mohamed El Nashaar, Professor of obstetric and gynecology Benha University, Benha University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: letrozole step-up protocol
Record Dates: First submitted 2017-06-07; First posted 2017-06-09 (Actual); Last update posted 2017-06-09 (Actual); Status verified 2017-06

CONDITIONS: Infertility Poly Cystic Ovary
MeSH Terms: interventions — Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Step Up group (Experimental): includes females taking Letrozole 5 mg tablets in a step-up protocol 5 mg in day one, 7.5 in day 2, 10 mg in days 3, 12.5 mg in day 4 and 15 in day 5 started in day 3 to day 7 of menstrual cycle.
  Interventions: Drug: Letrozole
- Control group (No Intervention): includes females taking Letrozole 5 mg tab orally once daily started in day 3 to day 7 of menstrual cycle.

INTERVENTIONS:
Drug: Letrozole — Letrozole is a third generation inhibitor that is emerging as a new oral agent for induction of ovulation.
  Arms: Step Up group

SUMMARY:
the aim of the study is to compare between the step-up and conventional protocols in ovulation induction in infertile women with PCOS

DETAILED DESCRIPTION:
The current study was conducted in private outpatient clinic after being approved by the medical ethics committee. The study is a prospective randomized study consisting of 90 Egyptian patients diagnosed as having infertility with pcos .

Sample size determination:

Group sample sizes of 42 and 42 achieve 80% power based on study finding carried out by (Galal et al., 2014) to detect a difference of 0.7 between the null hypothesis that both group means are 2.2 and the alternative hypothesis that the mean of group 2 is 1.5 with known group standard deviations of 1.5 and 0.6 and with a significance level (alpha) of 0.05000 using a two-sided Mann-Whitney test assuming that the actual distribution is uniform.

Sample size was calculated by PASS 11 Computer program for sample size calculation.

Taking into consideration 10% drop out rate, the sample size will be increased to 45 patients in group I and another 45 patients in group II.

Patients were divided into two groups with randomization sheet:

Group (I): includes 45 females taking Letrozole (old regimen).

Group (II): includes 45 females taking Letrozole 5 mg tab in a step-up protocol (new regimen).

ELIGIBILITY:
Inclusion Criteria:

* Age: 20 -37 years old.
* No conception for at least one year.
* Diagnosis of PCO as established by Rotterdam criteria, endometriosis diagnosed by laparoscope or unexplained infertility.

Exclusion Criteria:

* Age < 20 and > 35 years old.
* Uterine pathology e.g. fibroid or ovarian cyst.
* Hyperprolactinemia, hypo or hyperthyroidism.
* Impaired hepatic or renal function.
* History of hypersensitivity to study drugs.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2017-01-01 (Actual); Study Completion 2017-03-01 (Actual)

PRIMARY OUTCOMES:
Number of mature follicles | 2 weeks

SECONDARY OUTCOMES:
Pregnancy rate | one month

IPD SHARING:
Plan to Share IPD: Yes
Publish a manuscript